CLINICAL TRIAL: NCT02683161
Title: Pre to Postoperative Smoking Cessation
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Inability to adequately recruit participants during pre-post operative period.
Sponsor: Johns Hopkins University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB00071969
Record Dates: First submitted 2015-10-15; First posted 2016-02-17 (Estimated); Results first posted 2018-06-20 (Actual); Last update posted 2018-07-17 (Actual); Status verified 2018-06

CONDITIONS: Cigarette Smoking; Obesity
MeSH Terms: conditions — Cigarette Smoking; Obesity | interventions — Varenicline; Behavior Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Open-label trial (Other): All participants will attend approximately 6 study sessions pre-surgery and approximately 6 study sessions post-surgery, during which they will be provided three intervention components aimed at smoking cessation: a medication (varenicline) that has been FDA approved for smoking cessation, contingency management for biological evidence of nonsmoking, and behavioral counseling.
  Interventions: Drug: Varenicline; Behavioral: Contingency Management; Behavioral: Behavioral Counseling

INTERVENTIONS:
Drug: Varenicline — Varenicline will be administered as clinically indicated and will begin approximately 4-6 weeks prior to surgery. All participants will receive a 1-week dose induction period before transitioning to a full maintenance dose.
  Other Names: Chantix
Behavioral: Contingency Management — Contingency Management payments will begin on the target quit date (week 2) and will be in place for 5 weeks or until surgery (whichever is sooner). Participants will receive monetary incentives for biochemical evidence of smoking abstinence.
  Other Names: monetary incentives
Behavioral: Behavioral Counseling — All participants will complete a 3-session behavioral counseling intervention with a trained member of our study staff during 3 of the pre-surgical study visits. This brief counseling intervention provides participants with information about the experience of quitting smoking, including a benefits/disadvantage analysis, functional analysis of craving/risk periods, and skills-building exercises to prevent lapse and relapse.

SUMMARY:
The study will evaluate the feasibility of integrating an intensive pre- post-surgical smoking cessation intervention into a hospital setting, and assess measures of postsurgical recovery as a function of smoking cessation status.

DETAILED DESCRIPTION:
This study will evaluate the feasibility of integrating an intensive pre- post-surgical smoking cessation intervention (i.e., varenicline + monetary incentives + brief counseling) into a hospital setting by recruiting elective bariatric surgery patients and assessing theoretically relevant baseline characteristics (e.g., factors influencing smoking decisions, such as smoking motivation, delayed discounting, and distress tolerance) that may predict smoking cessation and post-surgical recovery outcomes. Participants will be required to attend a screening visit at the Behavioral Pharmacology Research Unit (BPRU) located on the Johns Hopkins Bayview Medical Campus, during which the participants will answer questionnaires, complete computerized tasks, and undergo sensory testing. Participants will then attend approximately 6 weekly study visits leading up to their bariatric surgery, and approximately 6 more weekly study visits after the surgery, as well as a 30-day follow-up visit, all located at the BPRU at Johns Hopkins Bayview. During the 6 pre-surgery visits and 6 post-surgery visits, participants will undergo an intensive smoking cessation treatment that includes administration of a medication called varenicline that has been FDA-approved for smoking cessation, as well as behavioral counseling sessions and monetary incentives for remaining smoke-free. After completing all study visits, participants will be asked to return for a 30-day follow-up visit, during which they will complete several study measures once more. Throughout the study, participants will be asked to periodically complete questionnaires, computerized tasks, and sensory testing. Investigators will also track outcomes associated with post-surgical recovery, including duration of hospital stay, hospital readmission, post-surgical complications, and prescription pain-killer use post-surgery.

ELIGIBILITY:
Inclusion Criteria:

* Smoker who has surgery scheduled 5-10 weeks in advance

Exclusion Criteria:

* being contraindicated for varenicline use
* evidence of psychiatric instability
* being unwilling/unable to adhere to the study schedule
* be unwilling to provide study access to medical records
* being otherwise judged by the study team to be inappropriate for study participation

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2015-10; Primary Completion 2017-07 (Actual); Study Completion 2017-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kelly E Dunn, Ph.D., Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins Bayview Medical Center, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No
The study was ended prematurely due to lack of recruitment. Data analysis is not possible and will not be reported.

RESULTS

PARTICIPANT FLOW:
Groups:
- Open-label Trial: Open label trial of varenicline, administered as clinically indicated, for smoking cessation in patients prior to and after surgery.
Period: Overall Study
Arm/Group | Open-label Trial
Started | 5
Completed | 5
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Open-label Trial
Number analyzed (Participants) | 5
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 5
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 4
  White | 1
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Change in Smoking Status
Description: Smoking abstinence is defined the change in number of self-reported cigarettes smoked per week
Time Frame: Assessed starting in week 2 of 12 weekly study visits
Measure: Mean (Standard Deviation); unit: Mean cigarettes per/day
Groups:
- Open-label Group: Participants received clinically-indicated dose of varenicline for smoking cessation.
Arm/Group | Open-label Group
Number analyzed (Participants) | 5
Mean cigarettes per/day
  Week 2 | 7.4 (4.1)
  Week 3 | 5.9 (2.3)
  Week 4 | 6.0 (2.1)
  Week 5 | 4.9 (1.3)
  Week 6 | 0.8 (0.7)
  Week 7 | 0 (0)
  Week 8 | 0 (0)
  Week 9 | 0 (0)
  Week 10 | 0.3 (0.6)
  Week 11 | 0 (0)
  Week 12 | 0 (0)

ADVERSE EVENTS:
Time Frame: 12-week open-label trial
Description: Adverse Event (AE) is defined as any event judged to be related to the medication and unexpected
Arm/Group | Open-label Trial
All-Cause Mortality (participants affected / at risk) | 0/5
Serious Adverse Events (participants affected / at risk) | 0/5
Other Adverse Events (participants affected / at risk) | 0/5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-09-07): https://cdn.clinicaltrials.gov/large-docs/61/NCT02683161/Prot_SAP_000.pdf